CLINICAL TRIAL: NCT07289607
Title: Effect of TECAR Therapy on Proprioception Function in Patients With Cervical Radiculopathy
Brief Title: Effect of TECAR on Cervical Radiculopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Ibrahim Ahmed Ibrahim Abu Ella, Lecturer, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005936
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cervical Radiculopathy
Keywords: TECAR , radiculopathy , Proprioception
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant
Masking Description: the patient in control group will receive sham TECAR therapy in addition to physical therapy exercise program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): Receives TECAR therapy in addition to standard physiotherapy.
  Interventions: Device: TECAR therapy
- Control group (Sham Comparator): Receives sham TECAR
  Interventions: Device: Sham TECAR therapy

INTERVENTIONS:
Device: TECAR therapy — TECAR Therapy A form of radiofrequency-based deep thermotherapy that delivers energy into tissues using frequencies between 300 kHz and 1.2 MHz.
  It heats from the inside out, giving deeper and more controlled thermal effects than superficial heat modalities.
  Arms: study group
Device: Sham TECAR therapy — TECAR Therapy a form of radiofrequency-based deep thermotherapy that delivers energy into tissues using frequencies between 300 kHz and 1.2 MHz.
  It heats from the inside out, giving deeper and more controlled thermal effects than superficial heat modalities.
  Arms: Control group

SUMMARY:
Cervical radiculopathy is characterized by pain, sensory disturbances, and impaired neuromuscular control due to nerve root compression. Proprioception dysfunction is often an overlooked component of this condition and can affect balance, posture, and motor control.

TECAR (Transfer of Energy Capacitive and Resistive) therapy is a form of deep heat electrotherapy known to improve tissue perfusion and neuromuscular function. Although TECAR is widely used for pain relief and mobility, its role in improving proprioception remains under-investigated, especially in cervical conditions. This study aims to bridge this gap by assessing proprioceptive outcomes in patients with cervical radiculopathy receiving TECAR therapy.

DETAILED DESCRIPTION:
* Design: Randomized controlled trial.
* Groups:
* Control group: Receives standard physiotherapy (e.g., cervical traction, exercises).
* Experimental group: Receives TECAR therapy in addition to standard physiotherapy.
* Duration: 3 sessions per week for 4 weeks.
* Outcome Measures: Joint position sense (JPS) using cervical repositioning tests, pain (VAS), functional disability (NDI).
* Assessment Times: Baseline and after 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosed cervical radiculopathy confirmed by clinical and radiological findings

  * Age 30-40 years
  * Pain duration > 4 weeks

Exclusion Criteria:

* • Cervical fracture or surgery

  * Vestibular disorders
  * Rheumatologic or neurological diseases
  * Cognitive impairment or pregnancy

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-05 (Estimated); Study Completion 2026-04-05 (Estimated)

PRIMARY OUTCOMES:
proprioception function | Baseline
  assessment of proprioception functions via CROM
Cervical ROM | Baseline
  ROM assessment via CROM

CONTACTS AND LOCATIONS:
Locations (1):
- Private Clinic, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
CONFIDENTIALITY OF THE RESEARCH

REFERENCES:
- [Background] Bameri A, Yassin M, Salehi R, Mansour Sohani S. The Effects of Manual Therapy with TECAR Therapy, on Pain, Disability and Range of Motion in Women with Non-specific Chronic Neck Pain. Med J Islam Repub Iran. 2024 Sep 17;38:107. doi: 10.47176/mjiri.38.107. eCollection 2024. PMID 39781327